CLINICAL TRIAL: NCT00423787
Title: Efficacy and Safety/Tolerability of Ragweed MATA MPL, a Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Efficacy and Safety/Tolerability of Ragweed MATA MPL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Head of Clinical Operations and Pharmacovigilance, Allergy Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RagweedMATAMPL301
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Allergoid; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity | interventions — ragweed MATA MPL

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ragweed MATA MPL (Experimental): modified Ragweed pollen allergen absorbed to Tyrosine and containing MPL adjuvant
  Interventions: Biological: Ragweed MATA MPL
- Placebo (Placebo Comparator): 4 injections of placebo 0.5 ml (2% tyrosine)
  Interventions: Biological: Ragweed MATA MPL

INTERVENTIONS:
Biological: Ragweed MATA MPL — 4 injections of increasing dose strength:
  1. 300 SU/0.5 ml
  2. 700 SU/0.5 ml
  3. 2000 SU/0.5 ml
  4. 6000 SU/0.5 ml

SUMMARY:
Ragweed MATAMPL has been developed by Allergy Therapeutics to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting ragweed pollens causing rhinitis and/or conjunctivitis with or without mild to moderate asthma bronchiale. The purpose of this study is to compare the efficacy of Ragweed MATAMPL versus placebo in ragweed-allergic subjects following 4 subcutaneous injections of study medication administered before the start of the 2007 ragweed pollen season

DETAILED DESCRIPTION:
Ragweed MATAMPL has been developed by Allergy Therapeutics to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting ragweed pollens causing rhinitis and/or conjunctivitis with or without mild to moderate asthma bronchiale.

An earlier formulation of Ragweed MATAMPL developed by Allergy Therapeutics (UK), Ltd, available commercially in Canada since the 1980's, is 'Pollinex®-R'. 'Pollinex®-R' is formulated with modified allergens (allergoids) of ragweed pollen extract adsorbed onto L tyrosine at 4% w/v. Related formulations developed by ATL, available commercially in selected European countries since the 1970´s on a Named Patient Basis, are 'Pollinex Tree', 'Pollinex Grass', 'Pollinex Quattro Trees' (previously known as MATA tree + MPL), and 'Pollinex Quattro Grass' (previously known as MATA grass + MPL).

Ragweed MATAMPL contains an extract of ragweed pollens. This extract is chemically modified with glutaraldehyde to produce the active ingredient, an allergoid. Such modification reduces the reactivity of the extract with IgE antibody. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivity is not seen. The modified extract is adsorbed to L-tyrosine as a depot formulation. MPL®, a purified, detoxified glycolipid derived from the cell walls of Salmonella minnesota, is also included in the current product formulation. This excipient/adjuvant is included to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to TH1-like T cell profile.

The current formulation is designed to provide a product that will be efficacious with only 4 injections, in contrast to the longer schedules currently in use with unmodified extracts. The product will also be safer to use than a formulation containing a similar mass of unmodified allergen extract as regards its ability to cause severe local allergic reactions or anaphylaxis, because of its reduced reactivity with IgE antibody. The modification is greater than 75%, so that only a small amount of unmodified allergen is remaining in the product.

The purpose of this study is to compare the efficacy of Ragweed MATAMPL versus placebo in ragweed-allergic subjects following 4 subcutaneous injections of study medication administered before the start of the 2007 ragweed pollen season.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent;
* Are 18 to 59 years of age;
* history of moderate to severe symptoms of seasonal allergic rhinitis and/or conjunctivitis ascribed to ragweed pollen exposure that required repeated use of antihistamines, nasal steroids, and/or leukotriene modifiers;
* history of moderate to severe symptoms in the past ragweed pollen season;
* positive skin prick test to ragweed pollen and a positive RAST or equivalent test to ragweed pollen;
* positive skin prick test to histamine;
* negative skin prick test to the negative control;
* forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted, with a FEV1/FVC ratio ≥ 70%;
* Women of childbearing potential must be using a medically acceptable method of birth control;
* able to understand and comply with study instructions;
* Demonstrate proper use of electronic diary with at least 85% compliance during the 1-week period between Visit 1 and Visit 2.

Exclusion Criteria:

* pregnant or lactating
* asthma requiring the daily use of controller medication;
* emergency room visit or admission for asthma in the 12 months prior to Visit 1;
* presence of secondary alteration at the affected organ (i.e., emphysema, bronchiectasis, nasal polyps, chronic sinusitis);
* auto-immune disease;
* acute or subacute (historic) atopic dermatitis, chronic dermatitis, urticaria factitia, and/or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of the skin prick test results;
* history or presence of diabetes, cancer or concomitant illness that, in the opinion of the Investigator, would pose a safety risk or compromise the interpretation of efficacy for this ragweed immunotherapy;
* history of angioedema;
* manifest pulmonary or cardiac insufficiency;
* current malignant disease;
* disorders of tyrosine metabolism (i.e., alcaptonuria, tyrosinemia);
* acute or chronic infection;
* any clinically significant abnormal laboratory value at Visit 1;
* Perennial Allergens: positive skin prick test at Visit 1 to: house dust mites, molds, or epithelia. In these cases, a careful history is to be taken and if moderate or severe symptoms are reported when exposed to the aforementioned allergens, the subject is to be excluded. Exception: the source of the allergen (cat, dog, horse) can be avoided for the entire study.
* Springtime Flowering Plant Allergens: positive skin prick test at Visit 1 to birch, oak, sycamore, ash, red maple, black walnut, American elm, or poplar. In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Exception: one or all of the listed allergens must not be tested if they are not common to the Investigator's region or, if common to the region, the treatment phase of the study can be initiated at least 30 days after the end of the allergen(s) season or treatment can be completed 30 days before the anticipated start of the allergen(s) season.
* Summertime Flowering Plant Allergens: positive skin prick test at Visit 1 to grass pollen mix or Bermuda grass. In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Exception: No testing is required if there is no overlap between grass / Bermuda grass and ragweed season and if treatment can be completed 30 days before the start of grass / Bermuda grass season. Bermuda grass must not be tested if it is not common to the Investigator's region.
* Late Summer/Autumn Flowering Plant Allergens: positive skin prick test at Visit 1 to: goosefoot/lamb's quarters, firebush/kochia, or English plantain. In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Exception: some or all of the listed allergens must not be tested if they are not common to the Investigator's region.
* Have inadequate washout period prior to screening (Visit 1). The following washout periods prior to Visit 1 are acceptable:

  * Oral or parenteral corticosteroids (1 month)
  * Inhaled, ocular or intranasal corticosteroids (1 day)
  * Mast cell stabilizers (7 days)
  * Intranasal or systemic decongestants including cold preparations (1 day)
  * Leukotriene modifiers (7 days)
  * Afrin (oxymetazoline hydrochloride) (14 days)
  * Antihistamines
* Once-daily or twice-daily antihistamines (7 days)
* Short-acting 3 or 4 times a day antihistamines (3 days)
* Hydroxyzine (14 days)

  * H2-blockers (1 day)
  * Other anti-inflammatory, anti-allergy, and any other medications which, in the opinion of the Investigator, may interfere with the study objectives should be considered on a case-by-case basis
  * Topical skin medications on the forearms (14 days);
* Require use of beta blockers;
* Are unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated);
* Have a history of anaphylactic reactions to foods, insect venom, exercise, or drugs;
* Have been treated with a preparation containing MPL® within 6 months prior to Visit 1;
* Have diseases with a pathogenesis interfering with the immune response, and who have received medication which could interfere with the results of the study;
* Have a history of allergy, hypersensitivity or intolerance to the excipients of the study medication;
* Have a history of allergy, hypersensitivity or intolerance to study relief medication;
* Have already undergone hyposensitisation therapy with comparable allergen extracts; An exception will be allowed if prior immunotherapy with comparable allergen was successful, symptoms reappeared some time after stopping the immunotherapy, and the immunotherapy was completed ≥ 3 years before Visit 1;
* Have participated in a clinical research trial with a new chemical substance within 4 weeks of Visit 1;
* Are unable or unwilling to cooperate with the Investigator and to comply with the protocol requirements, or not likely to complete the observation periods sufficiently;
* Have changed residence between geographical regions within the past 3 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 993 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of Ragweed MATA MPL versus placebo as measured by the combined allergy symptom (eyes and nose)+ medication scores self-reported by subjects during the 3 peak weeks of the 2007 ragweed pollen season. | 9 months

SECONDARY OUTCOMES:
Combined symptom + medication scores, Combined symptoms, Individual symptoms, Relief medication use, Specific immunological changes, quality of life, Health Assessments, Days absent from activities | 9 months
Adverse events, adverse reactions, clinical labs, ECG, and vitals | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl Jürgen Fischer von Weikersthal-Drachenberg, MD, Study Chair — Allergy Therapeutics
Locations (76):
- United States (59):
  - The Centre for Allergy, Asthma & Immunology, Waterbury, Connecticut
  - Allergy & Asthma Consultants, Atlanta, Georgia
  - Clinical Research Atlanta, Atlanta, Georgia
  - DataQuest Medical Research, Conyers, Georgia
  - Northeast Georgia Research Center LLC, Gainesville, Georgia
  - Allergy and Consultants, PC, Lilburn, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - University Consultants in Allergy/Immunlogy, Chicago, Illinois
  - Sneeze, Wheeze and Itch Associates, LLC, Normal, Illinois
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - Kansas City Allergy & Asthma, Overland, Kansas
  - Allergy & Arthritis Treatment Centre, Gardner, Massachusetts
  - Respiratory Medical Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute/West Health Building, Plymouth, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - Creighton University Medical Center Division of Allergy, Asthma and Immunology, Omaha, Nebraska
  - The Asthma and Allergy Centre, Papillion, Nebraska
  - Atlantic Research Center LLC, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Pulmonary & Allergy Associates, P.A., Summit, New Jersey
  - The Medical Center at Teaneck, Teaneck, New Jersey
  - AAIR Research Center, Rochester, New York
  - Ira Finegold, M.D., White Plains, New York
  - Regional Allergy & Asthma Consultants, Asheville, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Allergy & Asthma Care Centre, Fargo, North Dakota
  - Allergy & Respiratory Center, Canton, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Dr. Jeffrey Rosch Office and Research Centre, Altoona, Pennsylvania
  - Valley Clinical Research Centre, Easton, Pennsylvania
  - Allergy and Asthma Research of New Jersey Inc., Philadelphia, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Associates, Upland, Pennsylvania
  - Tricities Medical Research, Bristol, Tennessee
  - The Asthma Institute, PLLC, Chattanooga, Tennessee
  - The Allergy, Asthma & Sinus Centre PA, Knoxville, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Allergy & Asthma Associates Research Department, Austin, Texas
  - Lovelace Scientific Resources Allergy and Asthma Centre of Austin, Austin, Texas
  - AARA Research Centre, Dallas, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy & Asthma Associates, Houston, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Timber Lane Allergy & Asthma Research, South Burlington, Vermont
  - Commonwealth Clinic Research Specialists Inc., Richmond, Virginia
  - National Clinical Research, Richmond, Virginia
  - Allergy, Asthma & Sinus Centre, S.C., Greenfield, Wisconsin
  - Dean Foundation Medical Research, Madison, Wisconsin
  - University of Wisconsin, Madison, School of Medicine and Public Health, Madison, Wisconsin
  - Centre For Clinical Trials, Menomonee Falls, Wisconsin
  - Advanced Healthcare SC, Milwaukee, Wisconsin
  - Allergic Diseases SC, West Allis, Wisconsin
- Canada (17):
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Co-Medica Health Centre, Courtice, Ontario
  - McMaster University, Hamilton, Ontario
  - Kanata Allergy Services Ltd., Kanata, Ontario
  - Allied Research International Inc, Mississauga, Ontario
  - Alpha Medical Research Inc., Mississauga, Ontario
  - Niagara Clinical Research, Niagara Falls, Ontario
  - Northgate Medical Clinic, North Bay, Ontario
  - Allergy & Asthma Research Centre, Ottawa, Ontario
  - Melimar Allergy Laboratory Inc., Toronto, Ontario
  - Asthma, Allergy & Immunology, Toronto, Ontario
  - Gordon Sussman, 202 St. Clair Avenue West, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Omnispec Clinical Research, Mirabel, Quebec
  - Division of Clinical Immunology and Allergy, The McGill University Health Centre, Montreal, Quebec
  - Centre De Recherche Appliquée en Allergie De Quebec, Québec, Quebec
  - Q&T Research, Sherbrooke, Quebec